CLINICAL TRIAL: NCT01518192
Title: Risk Factors for Failure of Erythema Migrans Treatment - Comparison of Doxycycline and Cefuroxime Axetil for Treatment of Adult Patients With Erythema Migrans: Clinical and Microbiological Outcome.
Brief Title: Comparison of Doxycycline and Cefuroxime Axetil for Treatment of Erythema Migrans: Clinical and Microbiological Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Franc Strle, M.D., PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM-DC
Record Dates: First submitted 2010-06-28; First posted 2012-01-25 (Estimated); Results first posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2011-12

CONDITIONS: Erythema Migrans; Post-Lyme Disease Symptoms
Keywords: erythema migrans; doxycycline; cefuroxime axetil; post-Lyme disease symptoms; background symptoms in general population
MeSH Terms: conditions — Glossitis, Benign Migratory | interventions — Doxycycline; cefuroxime axetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1Doxycycline (Active Comparator)
  Interventions: Drug: doxycycline
- 2 Cefuroxime axetil (Active Comparator)
  Interventions: Drug: cefuroxime axetil

INTERVENTIONS:
Drug: doxycycline — 100 mg bid; 15 days
  Arms: 1Doxycycline
Drug: cefuroxime axetil — 500 mg bid; 15 days
  Arms: 2 Cefuroxime axetil

SUMMARY:
Background:

* While doxycycline is a standard antibiotic for treatment of erythema migrans in Europe as well as in the USA, the effectiveness of cefuroxime axetil in the treatment of adult patients with erythema migrans has been assessed only in the USA where the causative agent of Lyme disease is Borrelia burgdorferi, but not in Europe where the main etiologic agents are B. afzelii and B. garinii.
* Controversy exists over the significance and even the existence of post-Lyme disease symptoms because of the high rate of similar background symptoms in the general population.

Purpose:

The two main purposes of this European, prospective clinical trial in which doxycycline and cefuroxime axetil are compared in the treatment of adult patients with erythema migrans and which included a control group to address the significance of post-Lyme disease symptoms are:

* To assess and compare the effectiveness of doxycycline and cefuroxime axetil in the treatment of erythema migrans using clinical and bacteriological criteria (noninferiority testing approach), and
* to compare the frequency of post-Lyme disease symptoms in adult patients treated for EM with antibiotics and the frequency of similar symptoms in control subjects without Lyme disease.

DETAILED DESCRIPTION:
Sample size

Decisions were based on the following:

1. Number of patients with erythema migrans treated with doxycycline and cefuroxime axetil was determined assuming no difference in treatment outcome will be detected (non-inferiority testing).
2. The decision for a larger sample sizes than needed for 1. was done with the intention to evaluate the secondary outcome measure, i.e., to assess the difference between the frequency of new or increased symptoms in patients treated for early Lyme disease and the occurrence of the same symptoms in control subjects.

   1. We assumed that the outcomes in the two treatment groups will be comparable and that the patients could be combined for further analysis.
   2. To obtain a control group from the same geographical area, each patient was asked if she or he had a family member or friend who was within 5 years of her or his age and who was without a history of Lyme borreliosis. These persons were approached by a short written explanation of the investigation, containing also a request for their participation. We assumed that we will be able to get a corresponding control person not for all but for approximately 80-90% of patients.
   3. Under the assumption that approximately 15% of an estimated 200 patients would have new or increased symptoms at >6 months after enrollment into the study, a control group of 165 subjects would be sufficient to detect a >10 percentage point lower rate of new or increased symptoms in controls compared with patients at the 0.05 level (2-sided) with >90% power. To comply with drop outs at different time points we assessed that 280 patients and 230 controls should be included at baseline.

ELIGIBILITY:
Inclusion Criteria:

* patients 15 or more years old
* with typical erythema migrans
* evaluated between 6/06 and 9/06
* evaluated at the Lyme Disease Outpatient Clinic, University Medical Center Ljubljana, Slovenia.

Exclusion Criteria:

* history of Lyme disease in the past
* pregnancy
* lactation
* immunocompromising condition
* history of a serious adverse reaction to a beta-lactam or tetracycline drug
* receiving an antibiotic with known anti-borrelial activity within 10 days
* multiple erythema migrans lesions or an extracutaneous manifestation of Lyme disease.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daša Cerar, MD, Principal Investigator — Department of Infectious Diseases, University Medical Center Ljubljana, Ljubljana, Slovenia; Franc Strle, MD, Study Chair — Department of Infectious Diseases, University Medical Center Ljubljana, Ljubljana, Slovenia
Locations (2):
- Slovenia (2):
  - Institute of Microbiology and Immunology, Medical Faculty, University of Ljubljana, Ljubljana
  - Department of Infectious Diseases, University Medical Center Ljubljana, Ljubljana, Slovenia, Ljubljana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with typical erythema migrans, examined in the period from June to September 2006 at Lyme Disease Outpatient Clinic, University Medical Center Ljubljana, Slovenia
Pre-assignment Details: 113/398 patients were ineligible due to:
  * receiving antibiotic with known anti-borrelial activity (73)
  * multiple erythema migrans (16)
  * history of Lyme disease (12)
  * immunocompromising condition (4)
  * serious adverse reaction to study drugs (3)
  * pregnancy or lactation (4)
  * erythema migrans accompanied by meningitis (1)
Groups:
- Doxycycline: Patients were assigned to receive a 15-day oral treatment with doxycycline 100 mg twice daily.
  At baseline and at 14 days, 2, 6, and 12 months thereafter, patients were interviewed and examined. At baseline, a skin biopsy specimen was cultured; this procedure was repeated 2-3 months later in patients with a positive culture.
- Cefuroxime Axetil: Patients were assigned to receive a 15-day oral treatment with cefuroxime axetil 500 mg twice daily.
  At baseline and at 14 days, 2, 6, and 12 months thereafter, patients were interviewed and examined. At baseline, a skin biopsy specimen was cultured; this procedure was repeated 2-3 months later in patients with a positive culture.
- Controls: patients' family members or friends without a history of Lyme disease
Period: Overall Study
Arm/Group | Doxycycline | Cefuroxime Axetil | Controls
Started | 145 | 140 | 259
Completed | 116 | 114 | 224
Not Completed | 29 | 26 | 35
Not completed — Lost to Follow-up | 29 | 26 | 35

BASELINE CHARACTERISTICS:
Groups:
- Doxycycline; Cefuroxime Axetil: Patients were assigned to receive a 15-day oral treatment with either doxycycline 100 mg or cefuroxime axetil 500 mg twice daily, by alternating treatment regimens each week.
  Evaluations:
  At baseline and at 14 days, 2, 6, and 12 months thereafter, patients were interviewed and examined. At baseline, a skin biopsy specimen was cultured as previously described; this procedure was repeated 2-3 months later in patients with a positive culture.
- Controls: To obtain a control group from the same geographical area, each patient was asked if he/she had a family member or friend who was within 5 years of his/her age and had no history of Lyme disease (two of the potential control subjects were excluded due to this reason), and was not pregnant, lactating or immunocompromised.
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Cefuroxime Axetil | Controls | Total
Number analyzed (Participants) | 145 | 140 | 259 | 544
Age Continuous [Median (Full Range); unit: years] | 54 (14.6) [17 to 85] | 51.5 (14.9) [19 to 82] | 52 [15 to 85] | 52.5 (14.9) [15 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 77 | 125 | 286.0
  Male | 61 | 63 | 134 | 258.0
Region of Enrollment [Number; unit: participants]
  Slovenia | 145 | 140 | 259 | 544.0

OUTCOME MEASURES:

1. Primary Outcome: Objective Lyme Disease Manifestations and Post-Lyme Disease Symptoms at 14 Days
Description: Number of patients with objective manifestations of Lyme disease(persistence of erythema migrans or any of the extracutaneous-cardiac, nervous or skeletal-Lyme disease manifestations)and/or with post-Lyme disease symptoms in patients treated for solitary erythema migrans at 14 days post inclusion
Time Frame: at 14 days post inclusion
Population: All participants who followed the protocol were eligible for analysis
Measure: Number; unit: participants
Groups:
- Doxycycline: doxycycline 100 mg twice daily for 15 days
- Cefuroxime Axetil: cefuroxime axetil 500 mg twice daily for 15 days
Arm/Group | Doxycycline | Cefuroxime Axetil
Number analyzed (Participants) | 145 | 140
participants | 30 | 27

2. Secondary Outcome: New or Increased Symptoms Since Erythema Migrans in Patients and Controls at 6 Months.
Description: Comparison of the number patients and controls with new or increased symptoms since erythema migrans at 6 months.
Time Frame: 6 months
Population: all participants who followed the protocol
Measure: Number; unit: participants
Groups:
- Patients: patients with new or increased symptoms since erythema migrans at 6 months post inclusion
- Controls: controls with new or increased symptoms since enrollment at 6 months post inclusion
Arm/Group | Patients | Controls
Number analyzed (Participants) | 194 | 236
participants | 9 | 16

3. Primary Outcome: Adverse Events
Description: Number of patients reporting adverse events
Time Frame: at 14 days
Population: All participants who followed the protocol.
Measure: Number; unit: participants
Arm/Group | Doxycycline | Cefuroxime Axetil
Number analyzed (Participants) | 145 | 140
participants | 22 | 23

4. Primary Outcome: Objective Lyme Disease Manifestations and Post-Lyme Disease Symptoms at 2 Months
Description: Number of patients with objective Lyme disease manifestations and/or post-Lyme disease symptoms in patients treated for solitary erythema migrans at 2 months post inclusion
Time Frame: 2 months
Population: all participants who followed the protocol
Measure: Number; unit: participants
Arm/Group | Doxycycline | Cefuroxime Axetil
Number analyzed (Participants) | 136 | 134
participants | 19 | 14

5. Primary Outcome: Objective Lyme Disease Manifestations and Post-Lyme Disease Symptoms at 6months
Description: Number of patients with objective Lyme disease manifestations and/or post-Lyme disease symptoms in patients treated for solitary erythema migrans at 6 months post inclusion
Time Frame: 6 months
Population: all participants who followed the protocol
Measure: Number; unit: participants
Groups:
- Cefuroximew Axetil: cefuroxime axetil 500 mg twice daily for 15 days
Arm/Group | Doxycycline | Cefuroximew Axetil
Number analyzed (Participants) | 102 | 93
participants | 5 | 6

6. Primary Outcome: Objective Lyme Disease Manifestations and Post-Lyme Disease Symptoms at 12 Months
Description: Number of patients with objective Lyme disease manifestations and/or post-Lyme disease symptoms in patients treated for solitary erythema migrans at 12 months post inclusion
Time Frame: 12 months
Population: all participants who followed the protocol
Measure: Number; unit: participants
Arm/Group | Doxycycline | Cefuroxime Axetil
Number analyzed (Participants) | 116 | 114
participants | 3 | 4

7. Secondary Outcome: New or Increased Symptoms Since Erythema Migrans in Patients Controls at 12 Months.
Description: Comparison of the number of patients and controls with new or increased symptoms since erythema migrans at 12 months.
Time Frame: 12 months
Population: all participants who followed the protocol
Measure: Number; unit: participants
Groups:
- Patients: patients with new or increased symptoms since erythema migrans at 12 months post inclusion
- Controls: controls with new or increased symptoms since erythema migrans at 12 months post inclusion
Arm/Group | Patients | Controls
Number analyzed (Participants) | 230 | 224
participants | 5 | 21

8. Secondary Outcome: Selected Subjective Symptoms in Patients and Control Subjects
Description: Comparison of the number of patients and controls with selected 8 symptoms (fatigue, arthralgias, myalgias, headache, paresthesias, dizziness, irritability, or nausea) within the preceding week, irrespective of whether they were new or increased since erythema migrans.
Time Frame: Examination at 12 months
Population: all participants who followed the protocol
Measure: Number; unit: participants
Groups:
- Patients: patients with selected subjective symptoms at 12 months post inclusion
- Controls: controls with selected subjective symptoms at 12 months post inclusion
Arm/Group | Patients | Controls
Number analyzed (Participants) | 230 | 224
participants | 178 | 181

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Doxycycline | Cefuroxime Axetil | Controls
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/140 | 0/259
Other Adverse Events (participants affected / at risk) | 21/145 | 21/140 | 0/259
OTHER ADVERSE EVENTS (reported when occurring in more than 0.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=145) | Cefuroxime Axetil (N=140) | Controls (N=259)
Gastrointestinal symptoms (Gastrointestinal disorders) | 20 (20) | 21 (21) | 0 (0)
Photosensitivity (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Medical explanation besides Lyme disease of the symptoms in patients was based on history and physical examination, therefore some other medical explanations might have been missed. With regard to controls this was even more likely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No